CLINICAL TRIAL: NCT05762588
Title: JuggerKnot With BroadBand Tape Post Market Clinical Follow-Up Study
Brief Title: JuggerKnot With Broadband PMCF Study
Status: Active, not recruiting | Type: Observational
Sponsor: Riverpoint Medical (Industry)
Responsible Party: Sponsor
Other Study IDs: JUGGPMCF
Record Dates: First submitted 2023-02-27; First posted 2023-03-09 (Actual); Last update posted 2025-08-17 (Actual); Status verified 2025-08

CONDITIONS: Shoulder Injuries; Hip Injuries; Foot Injury; Ankle Injuries; Knee Injuries
Keywords: Soft tissue fixation
MeSH Terms: conditions — Shoulder Injuries; Hip Injuries; Foot Injuries; Ankle Injuries; Knee Injuries

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- Patients requiring soft tissue fixation of the shoulder, knee, foot/ankle, elbow, or hip
  Interventions: Device: Juggerknot with Broadband tape

INTERVENTIONS:
Device: Juggerknot with Broadband tape — The JuggerKnot system is comprised of a coreless sleeve structure and suture. The anchors are intended for use in soft tissue to bone fixation by bunching against the bone when deployed. The anchor sleeve material is polyester. Suture materials are ultra-high molecular weight polyethylene. The device has 510K FDA clearance.

SUMMARY:
The purpose of the study is to collect post-market clinical follow-up data, which is needed to confirm the safety and performance of the JuggerKnot device and meet existing EU regulatory requirements.

ELIGIBILITY:
Inclusion Criteria:

1. Undergoing soft tissue fixation of the shoulder, knee, foot/ankle, elbow, or hip where the JuggerKnot with BroadBand anchor is indicated;
2. Male or non-pregnant female ≥ 18 years of age;
3. Willing to provide informed consent and comply with the required follow-up period.

Exclusion Criteria:

1. Infection where implantation of the device would be compromised;
2. Conditions including blood supply limitations and insufficient quantity or quality of bone or soft tissue;
3. Known allergy to one of the JuggerKnot with BroadBand components;
4. Mental or neurologic conditions who are unwilling or incapable of following postoperative care instructions or patients who are otherwise unwilling or incapable of doing so.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Approximately 30 participants at approximately 3 clinical sites in the United Sates are planned to be enrolled.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2023-11-30 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Clinical Success | 6 months
  Defined as freedom from reintervention due to JuggerKnot with BroadBand failure. Absence of device migration loosening or pull-out.

SECONDARY OUTCOMES:
Technical and Procedural Success | Intraoperatively
  Successful bone to soft tissue fixation without complications such as anchor pull-out, suture breakage or suture pull through.
PROMIS Physical Function Score | Change from baseline to 6 months
  The PROMIS Global-10 is a 10-item patient-reported questionnaire in which the response options are presented as 5-point (as well as a single 11-point) rating scales. The results of the questions are used to calculate two summary scores: a Global Physical Health Score and a Global Mental Health score. These scores are then standardized to the general population, using the "T-Score".
VAS Pain Score | Change from baseline to 6 months
  A VAS consists of a line, often 10 cm long, with verbal anchors at either end, similar to an NRS (e.g., "no pain" on the far left and "the most intense pain imaginable" on the far right). The patient places a mark at a point on the line corresponding to the patient's rating of pain intensity.
Change in degrees of Range of Motion (ROM) measured by Goniometer | Change from baseline to 6 months
  The extent or limit to which a part of the body can be moved around a joint or a fixed point. ROM will depend on the anatomy being studies. ROM will be measured by goniometer.

CONTACTS AND LOCATIONS:
Locations (1):
- MedStar Health Research Institute, Hyattsville, Maryland, United States

IPD SHARING:
Plan to Share IPD: No